CLINICAL TRIAL: NCT02440646
Title: The Natural History of Coronary Atherosclerosis Within the Concept of the Glagovian Arterial Remodeling in REAL-world Stable Chest Pain Population Who Underwent nonInvasive compuTed tomographY Angiography in Comparison With Invasive Quantitative Coronary Angiography and Multimodality Imaging Handled by the Advanced Post-processing Software: Clinical potentIal and Safety
Brief Title: Natural History of Coronary Atherosclerosis in Real-World Stable Chest Pain Patients Underwent Computed Tomography Angiography in Comparison With Invasive Multimodality Imaging
Acronym: REALITY
Status: Terminated | Type: Observational
Why Stopped: The study is terminated due to cessation of the research collaboration with Russian institutions
Sponsor: Central Clinical Hospital of the Russian Academy of Sciences (Other Government)
Collaborators: Ural State Medical University (Other); De Haar Research Task Force (Industry); Center of Endosurgery and Lithotripsy, Moscow, Russia (Other); JHWH International Advanced Cardiovascular Imaging Consortium (Unknown); Medis Medical Imaging Systems B.V. (Unknown); Pie Medical Imaging B.V. (Unknown); De Haar Research Foundation (Other)
Responsible Party: Principal Investigator, Alexander Kharlamov, MD, FESC, FACC, FEACVI, Principal investigator and coordinator of the REALITY project, De Haar Research Task Force
Other Study IDs: REALITY Advanced
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Coronary Atherosclerosis; Coronary Artery Disease; Contrast-induced Nephropathy; Cerebrovascular Disease; Alzheimer Disease; Chronic Coronary Insufficiency; Stable Chronic Angina
Keywords: Computed tomography angiography; Quantitative coronary angiography; Coronary artery disease; Natural history of atherosclerosis; Radiocontrast-induced thyroid dysfunction; Contrast-induced nephropathy; Plaque burden; Glagovian artery remodeling; Radiation dose; SYNTAX score; Fractional flow reserve; Optical coherence tomography; Intravascular ultrasound; Intravascular imaging; Cardiac magnetic resonance; Echocardiography; Single photon emission computed tomography
MeSH Terms: conditions — Coronary Artery Disease; Cerebrovascular Disorders; Alzheimer Disease; Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood samples to test the main hypothesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CCTA group: All stable chest pain comers admitted to the chest-pain outpatient or inpatient cardiac center with the chronic coronary syndrome who underwent functional tests (CMR and/ or SPECT, and Echo are mandatory) and coronary computed tomography angiography (CCTA) without further immediate quantitative coronary angiography (QCA), applicable intravascular imaging (FFR, QFR, OCT, IVUS, VH-IVUS) and/ or percutaneous intervention (PCI).
  Interventions: Radiation: Coronary computed tomography angiography
- CCTA + Invasive group: All stable chest pain comers admitted to the chest-pain outpatient or inpatient cardiac center with the chronic coronary syndrome who underwent functional tests (CMR, and/ or SPECT, and Echo are mandatory) and coronary computed tomography angiography (CCTA) with further quantitative coronary angiography (QCA), applicable intravascular imaging (FFR, QFR, OCT, IVUS, VH-IVUS) with or without implantation of a stent.
  Interventions: Radiation: Quantitative coronary angiography, intravascular imaging with percutaneous intervention

INTERVENTIONS:
Radiation: Coronary computed tomography angiography — The coronary arteries will be visualized with the MSCT scan CT 5000 Ingenuity (Philips, The Netherlands) or systems from any other vendors.
  Other Names: CCTA
  Groups: CCTA group
Radiation: Quantitative coronary angiography, intravascular imaging with percutaneous intervention — Coronaries will be shot with Artis zee (Siemens, Germany) or systems from any other vendors. In case if necessary the procedure will be delayed for intravascular imaging (FFR, QFR, OCT, IVUS, VH-IVUS) and/ or percutaneous intervention (with implantation of the medical device).
  Other Names: QCA; Coronary intravascular imaging
  Groups: CCTA + Invasive group

SUMMARY:
In a prospective international multicenter observational study, 1080 stable chest pain patients (REALITY Advanced registry of CCTA patients) with the suspected chronic coronary syndrome will be enrolled. All of them will undergo computed tomography angiography, CMR and/ or SPECT, and Echo. One of the cohorts will be examined with multimodality invasive imaging including quantitative coronary angiography, FFR, QFR with or without further percutaneous coronary intervention, OCT, and some of them - with IVUS, VH-IVUS. The plaque size and relevant stenosis, a composition of the atherosclerotic lesion, major adverse cardiovascular events (all-cause death, death from cardiac causes, myocardial infarction, or rehospitalization due to unstable or progressive angina, ischemia-driven revascularization) will be judged to be related to either originally treated (culprit) lesions or untreated (non-culprit) lesions. Moreover, the clinical potential of both non-invasive and invasive imaging, as well as anatomical vs functional modalities in two real-world patient flows, will be estimated with the special focus on the natural progression of atherosclerosis, clinical outcomes, and safety (contrast-induced nephropathy, radiocontrast-induced thyroid dysfunction, and radiation dose). The diagnostic accuracy will be analyzed.

The follow-up period will achieve 12 months prospectively with collected clinical events and imaging outcomes which will be determined at the baseline and 12-month follow-up.

The independent ethics expertise will be provided by the Ural State Medical University (Yekaterinburg, Russia) and Central Clinical Hospital of the Russian Academy of Sciences (Moscow, Russia). The monitoring of the clinical data with imaging as well as further CoreLab expertise (expert-level post-processing multimodal imaging software of Medis Imaging B.V., Leiden, The Netherlands) will be provided by De Haar Research Task Force, Amsterdam-Rotterdam, the Netherlands. FFR-CT is scheduled to be assessed by the ElucidVivo Research Edition software from Elucid Bio, Boston, MA, U.S.A.

The REALITY project is a part of the JHWH (Jahweh) International Advanced Cardiovascular Imaging Consortium. The main objective of the Consortium that is uniting international efforts of both Academia and Industry is a synergistic development of the advanced machine-learning imaging software in order to integrate benefits of both non-invasive and invasive imaging providing the daily clinical practice with the robust tool for the anatomical and functional examination of coronary atherosclerosis, PCI-related arterial remodeling, and relevant myocardial function.

DETAILED DESCRIPTION:
Invasive coronary angiography with fractional flow reserve (FFR) is considered as the reference standard of daily clinical practice. This invasive approach is associated with potentially life-threatening complications, high expenditures, relatively high radiation exposure, and some patient discomfort. Noninvasive cardiac computed tomography angiography (CCTA) becomes a robust alternative to the invasive approach, especially when supported by other functional and anatomical noninvasive imaging modalities such as cardiac magnetic resonance (CMR), single-photon emission computed tomography (SPECT), and echocardiography (Echo). Notwithstanding, their invasive counterpart, particularly a multimodal intravascular imaging (including fractional flow reserve/ FFR, quantitative flow reserve/ QFR, optical coherence tomography/ OCT, intravascular ultrasound/ IVUS, VH-IVUS) is able to rule out the high-risk, vulnerable and obstructive atherosclerosis dramatically optimizing clinical outcomes. The clinical value of these techniques remains questionable, especially if compared between noninvasive and invasive imaging methods.

The modern-day imaging modalities allow clinical cardiology to study the natural history of atherosclerosis that can predict certain clinical outcomes paving the way for a reduction of cardiovascular mortality. The retrospective studies have shown that most atherosclerotic plaques responsible for future acute coronary syndromes are angiographically mild, and the lesion-related risk factors for major adverse cardiovascular events (MACE) are poorly understood. Pathological studies have shown that thrombotic coronary occlusion after rupture of a lipid-rich atheroma with only a thin fibrous layer of intimal tissue covering the necrotic core (a thin-cap fibroatheroma) is the most common cause of myocardial infarction and death from cardiac causes. However, the prospective identification of thin-cap fibroatheromas has not been achieved, in part because the imaging tools to identify them in vivo did not exist until recently (Stone GW, et al, 2011; DOI: 10.1056/NEJMoa1002358). Both CCTA and quantitative coronary angiography (QCA) provide us with the potential of the advanced imaging of atherosclerotic lesions, but accuracy and safety remain the keystone limitations of these approaches. CCTA has the unique advantage over detecting non-calcifying plaques in addition to calcifying lesions, thus allowing for direct visualization of early atherosclerosis stages such as lipid and fibrous atheroma, which are risk factors for future coronary events. Long-term studies report an increased risk of the adverse outcomes associated with vulnerable fibroatheroma, whereas calcifying lesions tend to remain rather stable. Studies investigating the accuracy, outcome, and, thus, the diagnostic benefit of coronary CCTA in chest pain patients are scarce (Plank F, et al, 2014; doi:10.1136/openhrt-2014-000096). The accuracy of some advanced imaging modalities has recently developed to overcome existing limitations, however, the accuracy and precision of those measurements in the different stage lesions have not been established (Kan J, et al, 2014).

In a prospective international multicenter observational study, 1080 stable chest pain patients (REALITY Advanced registry of CCTA patients) with the suspected chronic coronary syndrome will be enrolled. All of them will undergo computed tomography angiography, CMR, and/ or SPECT, and Echo. One of the cohorts will be examined with multimodality invasive imaging including quantitative coronary angiography with or without further percutaneous coronary intervention, FFR, QFR, OCT, and some of them - with IVUS, VH-IVUS. The plaque size and relevant stenosis, a composition of the atherosclerotic lesion, major adverse cardiovascular events (all-cause death, death from cardiac causes, myocardial infarction, or rehospitalization due to unstable or progressive angina, ischemia-driven revascularization) will be judged to be related to either originally treated (culprit) lesions or untreated (non-culprit) lesions. Moreover, the clinical potential of both non-invasive and invasive imaging, as well as anatomical vs functional modalities in two real-world patient flows, will be estimated with the special focus on the natural progression of atherosclerosis, clinical outcomes, and safety (contrast-induced nephropathy, radiocontrast-induced thyroid dysfunction, and radiation dose). The diagnostic accuracy will be analyzed.

The follow-up period will achieve 12 months prospectively with collected clinical events and imaging outcomes which will be determined at the baseline and 12-month follow-up.

The independent ethics expertise will be provided by the Ural State Medical University (Yekaterinburg, Russia) and Central Clinical Hospital of the Russian Academy of Sciences (Moscow, Russia). The monitoring of the clinical data with imaging as well as further CoreLab expertise (expert-level post-processing multimodal imaging software of Medis Imaging B.V., Leiden, The Netherlands) will be provided by De Haar Research Task Force, Amsterdam-Rotterdam, the Netherlands.

The clinical data of the REALITY Advanced Registry include information of the complex examination with a 64-128-slice CT, two interviews with the risk factor modification recommendations, lab screening (serum fasting glucose, asparagine transaminase, alanine transaminase, total bilirubin, carbamide/ urea, creatinine, total cholesterol, triglycerides, LDL cholesterol, HDL cholesterol, VLDL cholesterol), markers of the myocardium damage (myoglobin, troponin I, creatine kinase, creatine kinase-MB, brain natriuretic peptide - NT-proBNP), complete blood count, ECG, and Echo. The Registry patients will be tested with HeartAge, SCORE, Duke ACC/ AHA, Duke - DCS, Diamond-Forrester - DFM, The Seattle Angina Questionnaire - SAQ, Duke Activity Status Index -DASI, and EQ-5D-5L. Patients will be screened for the major risk factors and their modification: unhealthy blood cholesterol levels, high blood pressure, smoking, insulin resistance, diabetes, overweight or obesity, lack of physical activity, unhealthy diet (elements of Mediterranean and so-called 'Russian' diet), older age, genetic or lifestyle factors, family history of early heart disease. Moreover, such factors as CRP, sleep apnea, stress, and alcohol consumption will be assessed.

The eligibility criteria which the candidates must have fulfilled will be verified and the optimal clinical strategy will be estimated by the Heart Team, the Data Safety, and Monitoring Board. The clinical outcomes will be examined by the independent clinical endpoint adjudication committee.

The CCTA will be undergone in accordance with the 2016 SCCT (Society of Cardiovascular Computed Tomography) guidelines for the performance and acquisition of coronary computed tomographic angiography (Journal of Cardiovascular Computed Tomography/JCCT 2016;10:435e449). The results of the CCTA will be interpreted taking into account the 2020 SCCT Expert Consensus Document on Coronary CT Imaging of Atherosclerotic Plaque (JCCT 2020) and the 2021 SCCT Expert Consensus Document on Coronary Computed Tomographic Angiography (JCCT 2021). All non-invasive and invasive imaging procedures will be performed in accordance with local site practice, national, international, and societal guidelines including Society for Cardiovascular Magnetic Resonance (SCMR), American Society of Echocardiography (ASE), European Association of Percutaneous Cardiovascular Interventions (EuroPCR/ EAPCI), Society for Cardiovascular Angiography and Interventions (SCAI).

The imaging data from non-invasive (CCTA, FFR-CT, CMR, SPECT, Echo) and invasive (QCA, FFR, QFR, OCT, IVUS, VH-IVUS) methods will be handled and analyzed with the expert-level post-processing imaging software (Medis Suite Solutions: MR, XA, QFR, CT, Intravascular, Ultrasound) from Medis Medical Imaging Systems B.V. (Leiden, The Netherlands), if applicable. Raw imaging data will be transferred to the independent CoreLab (De Haar Research Task Force, Rotterdam-Amsterdam, The Netherlands) and analyzed by two experienced readers, blinded to the patient's information. The interobserver disagreements will be resolved by a third reader. FFR-CT is scheduled to be assessed by the ElucidVivo Research Edition software from Elucid Bio, Boston, MA, U.S.A.

The REALITY project is a part of the JHWH (Jahweh) International Advanced Cardiovascular Imaging Consortium. The main objective of the Consortium that is uniting international efforts of both Academia and Industry is a synergistic development of the advanced machine-learning imaging software in order to integrate benefits of both non-invasive and invasive imaging providing the daily clinical practice with the robust tool for the anatomical and functional examination of coronary atherosclerosis, PCI-related arterial remodeling, and relevant myocardial function.

The main aim of the REALITY Advanced trial is to evaluate the natural history of atherosclerosis within the concept of the Glagovian arterial remodeling in stable chest pain patients with the assessment of the clinical potential/ prognostic value and safety of the different noninvasive and invasive imaging tools as CCTA (and/ or CMR, SPECT, Echo), QCA, FFR, QFR, and applicable intravascular imaging (OCT, IVUS, VH-IVUS) handled with the advanced post-processing imaging software. Some preventive and therapeutic strategies will be examined, focusing on the place in routine clinical practice of such noninvasive imaging approach as CCTA vs relevant invasive imaging. The currently developed noninvasive imaging tools, including 64-128-320-slice CCTA processed with the high-accuracy machine-learning imaging software, can upgrade the noninvasive imaging's clinical value in contrary to the invasive approach, evaluating the significance of coronary atherosclerosis with related high-risk features of the arterial remodeling, predicting clinical outcomes, and avoiding unnecessary invasive intravascular interventions. The optimization of the diagnostic strategy and associated interventional approach can pave the way for dramatic improvement of clinical outcomes and cost-effectiveness of coronary artery disease (CAD) clinical management and, therefore, for substantial cardiovascular mortality reduction.

The REALITY Advanced trial pursued several objectives as follows:

1. To compare anatomical methods of noninvasive (CCTA, CMR) vs. invasive (QCA, OCT, IVUS, VH-IVUS) imaging with a focus on the options such as:

   1. High-risk and vulnerable features of lesions, including plaque composition with particular attention to the size of the necrotic core, the thickness and histological condition of the cap, signs of erosion, rupture, local thrombosis,
   2. Arterial remodeling,
   3. Significance of a 40% plaque burden as a keystone threshold for progression of atherosclerosis and clinical outcomes,
   4. Perivascular inflammation,
   5. Culprit vs. non-culprit lesions,
   6. Assessment of the blood flow physiological patterns, including invasively measured vs. calculated fractional flow reserve, wall shear stress (if applicable) derived from both noninvasive and invasive imaging and handled by the advanced post-processing imaging software,
   7. Diagnostic accuracy in comparison between various imaging modalities.
2. To match noninvasive and invasive anatomical (CCTA, QCA, OCT, IVUS, VH-IVUS) vs. functional (Echo, CMR, SPECT, MSCT) imaging, particularly if the anatomical significance of coronary atherosclerosis compared to the time trajectory of the cardiac function with a focus on:

   1. Ischemia (assessed by stress testing with CMR, SPECT, MSCT, Echo),
   2. Strain (both regional and global with different imaging modalities),
   3. Inflammation, including edema, fibrosis, particularly with CMR (hyperemia with EGE/ early gadolinium enhancement, edema with T2 weighted imaging, and scar/necrosis or fibrosis with LGE/ late gadolinium enhancement),
   4. Local coronary hemodynamics,
   5. Diagnostic accuracy in comparison between various imaging modalities.
3. To calculate the predictive value (with some risk stratification models) of different noninvasive and invasive imaging modalities amid various therapeutic strategies and invasive interventions. The performance of each strategy will be examined for sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and receiver operator characteristic (ROC) curve.
4. To conduct epidemiological analysis of the involved population and evaluate the cost-effectiveness of the different noninvasive and invasive strategies in stable chest pain patients, including:

   1. Direct effects: cost of imaging test, cost of complications due to imaging testing, effects of radiation, effects of contrast material, other complications of noninvasive and invasive imaging, psychological effects of the imaging test,
   2. Indirect effects: cost of the treatment, cost of complications of treatment, cost of health outcome, medical pathway, and health outcome depending on a medical decision based on the image test result, psychological effects of the test result.

ELIGIBILITY:
Inclusion Criteria:

* all stable chest pain comers with chronic coronary syndrome or angina equivalent consistent with the manifestation of the stable coronary artery disease (by the 2019 Guidelines on Chronic Coronary Syndrome);
* age between 40 and 79 years old;
* patient must have one or two-vessel disease in a native coronary vessel requiring or not requiring PCI without indications for immediate bypass surgery with any SYNTAX score;
* lesions may be either de novo or restenotic;
* successful, uncomplicated PCI could be performed in the culprit vessels and all culprit lesions, but there should be no events or complications between the procedures of PCI in the past and six months before admission to the Chest Pain Center;
* the non-culprit vessel should have no flow-limiting lesions (but any plaque burden) and be available for imaging. The non-culprit vessel must be considered safe for imaging evaluation;

Exclusion Criteria:

* any acute comorbidities;
* patient has had a documented ST-elevation acute myocardial infarction within the 24 hours or acute coronary syndrome (unstable angina, myocardial infarction) during four weeks before admission to the Chest Pain Center;
* patient has had a recent PCI (last 6 months before admission to the Chest Pain Center) unless the patient is undergoing a staged procedure for dual vessel treatment;
* unprotected left main lesion location;
* imaging evidence of severe calcification (CCTA calcium scoring with a CAC>1000) or marked tortuosity of the vessel;
* culprit lesion is located within or distal to an arterial or saphenous vein graft;
* untreated, significant coronary lesion with a >50-75% diameter stenosis remaining in the culprit vessel after the planned intervention (branch stenosis is permitted) unless allowed by the Heart Team, or the Institutional Review Board (IRB), or the Data Safety and Monitoring Board (DSMB);
* lesion or vessel contains visible thrombus within the imaging procedure;
* patient has an additional lesion that requires intervention within 180 days after the initial hospitalization unless allowed by the Heart Team, or the IRB, or the DSMB;
* any diameter stenosis more than 75% in the non-culprit vessel;
* indications for immediate bypass surgery within one year of enrollment with the SYNTAX above 34 (including multi-vessel disease requiring intervention in all three major coronary arteries);
* decompensated hypotension or heart failure requiring intubation, inotropes, intravenous diuretics, or intra-aortic balloon counterpulsation (including the presence of cardiogenic shock);
* patient has a known left ventricular ejection fraction <40% or history of decompensated congestive heart failure;
* uncontrolled tachycardia or refractory ventricular arrhythmia;
* presence of cardiac implants;
* acute conduction system disease requiring a pacemaker;
* uncontrolled hypokalemia or digitalis intoxication;
* uncontrolled arterial hypertension;
* moderate or severe pulmonary hypertension with pulmonary artery systolic pressure >35 mmHg;
* severe disorders of blood coagulation system/ coagulopathy;
* fever; active infective endocarditis; active COVID-19 infection; any active or severe chronic viral infections; sepsis;
* HIV infection: CDC acute retroviral syndrome/ acute HIV infection, CDC stage 3/ WHO stage 4 (AIDS; the CD4+ cell count is less than 200 or the percent of CD4+ cells is less than 15% of all lymphocytes); however, the subjects of the HIVE trial (NCT04810364) are allowed, but with chronic HIV infection (CDC stages 1, 2/ WHO stages 1, 2, 3) only;
* tuberculosis;
* creatinine clearance with GFR of <45 mL/min/1.73 m2 (severe CKD, G3b-G4-G5) by CKD-EPI (2009) or <45 mL/min by Cockroft-Gault (1976); a few reasons are there for these limitations, a) many medications are contraindicated and/ or dosages must be decreased in patients with severe CKD, b) already-in-use metformin with eGFR ≥45 mL/min/1.73 m2 is not an exclusion criterion, and metformin must be not stopped at the time of or before studies with IV contrast or withheld for 48 hours after the procedure, c) to reduce contrast material and radiation dose and therefore to prevent contrast-associated acute kidney injury, all the procedures with intravascular contrast (CCTA, CMR, SPECT, coronary angiography and any related invasive intravascular procedures) cannot be performed altogether subsequently during 24-48 hours, but it must undergo within two weeks with the recommended minimum break time between procedures of 48 hours and proper preventive hydration of the recruited patients.
* need for dialysis;
* liver cirrhosis;
* severe endocrine disorders (diabetes is permitted) including pre-existing thyroid diseases unless allowed by the Heart Team, or the IRB, or the DSMB;
* patient has a known hypersensitivity, allergy, or contraindication to any of the following: aspirin, heparin, clopidogrel, and ticlopidine, or to contrast (including iodine and gadolinium) that cannot be adequately pre-medicated;
* severe asthma or chronic obstructive pulmonary disease with FEV-1 below 50%;
* patient has other severe medical illness or recent history of substance abuse that may cause non-compliance; confound the data interpretation or is associated with an anticipated limited life expectancy of less than one year;
* stage IV cancer;
* patient on the transplant waiting list;
* moderate and severe anemia with hemoglobin below 11.0 g/dL, any severe blood diseases;
* acute or recent history of gastrointestinal bleeding;
* pregnancy;
* stroke or CVA within three months before admission to the Chest Pain Center;
* mental diseases, claustrophobia, inability for patient cooperation;
* prior participation in this study or patient is currently enrolled in another investigational use device, imaging, or drug study that has not been reached its primary endpoint.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All stable chest pain comers with a chronic coronary syndrome without acute angina who underwent CCTA (CMR, and/ or SPECT, and Echo are mandatory) and/ or QCA, applicable intravascular imaging (OCT, IVUS, VH-IVUS) with or without further PCI.
Sampling Method: Probability Sample
Enrollment: 1080 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Change of per cent of plaque burden from baseline to follow-up as assessed by either CCTA or QCA | At 12 months after the baseline imaging procedure
  Plaque burden for both culprit and non-culprit lesions will be calculated as a lesion volume (vessel volume-lumen volume)/lumen volume x 100. The variable will be adjusted for computed tomography angiography (CCTA) and quantitative coronary angiography (QCA) including the available methods of both noninvasive (CMR, SPECT) and invasive (OCT, IVUS, VH-IVUS) imaging.
Number of participants with major adverse cardiac events that are related to plaque burden | At 12 months after the baseline imaging procedure
  The composite of cardiac death, cardiac arrest, myocardial infarction, acute coronary syndrome, revascularization by coronary artery bypass surgery (CABG) or percutaneous coronary intervention (PCI), or rehospitalization for angina for patients with both culprit- and non-culprit-lesion-related events. Event rates will be determined at: hospital, at 12 months. The results will be compared with the CCTA-related predictive model of the ElucidVivo Research Edition software from Elucid Bio, Boston, MA, U.S.A.
Head-to-head comparison between non-invasive (CCTA, FFR-CT, CMR, SPECT, Echo) and invasive imaging (QCA, FFR, QFR, OCT, IVUS, VH-IVUS) | At baseline and 12 months after the baseline imaging procedure
  A comparison will be performed to assess the diagnostic accuracy of both noninvasive and invasive imaging approaches for the detection of obstructive coronary artery disease, comprehensive characterization of atherosclerosis. The imaging data will be analyzed by the expert-level post-processing software.
Non-invasive imaging for risk stratification | At 12 months after the baseline imaging procedure
  To determine the prognostic value of CCTA, CMR, SPECT, and Echo handled with the expert-level post-processing software for predicting cardiac death and nonfatal myocardial infarction. The results will be compared with the CCTA-related predictive model of the ElucidVivo Research Edition software from Elucid Bio, Boston, MA, U.S.A.
Invasive imaging for risk stratification | At 12 months after the baseline imaging procedure
  To determine the prognostic value of QCA, FFR, QFR, OCT, IVUS, VH-IVUS, handled with the expert-level post-processing software for predicting cardiac death and nonfatal myocardial infarction. The results will be compared with the CCTA-related predictive model of the ElucidVivo Research Edition software from Elucid Bio, Boston, MA, U.S.A.
Diagnostic accuracy of non-invasive and invasive imaging | At baseline and 12 months after the baseline imaging procedure
  Determining the diagnostic accuracy of stand-alone cardiac imaging modalities including CCTA, CMR, SPECT, Echo, QCA, FFR, QFR, OCT, IVUS, VH-IVUS.
Progression of atherosclerosis and plaque composition in comparison between non-invasive and invasive imaging methods | At baseline and 12 months after the baseline imaging procedure
  The progression of atherosclerosis will be quantitatively characterized by the parameters of the lesions (e.g. plaque burden, cap thickness, arterial remodeling, presence of erosions or rupture, malaposition of stent, a vessel injury score and so on). The imaging data will be handled with the expert-level post-processing software.
Comparison between anatomical and functional imaging modalities | At baseline and 12 months after the baseline imaging procedure
  The anatomical (CCTA, CMR, SPECT, QCA, OCT, IVUS, VH-IVUS) and functional (MSCT, CMR, SPECT, Echo, FFR-CT, FFR, QFR) imaging modalities will be compared to assess the difference between the progression of coronary atherosclerosis, condition of blood flow, and myocardial function in the field of interest. The myocardium will be visualized with the CMR system Ingenia 3.0T (Philips, The Netherlands) or systems from any other vendors.

SECONDARY OUTCOMES:
Change of serologic markers of inflammation from baseline to follow-up that are related to cardiovascular events and intervention | At baseline and 12 months after the baseline imaging procedure
  Variables will be evaluated for predictive value relative to recurrent events in mmol/L.
Number of participants with procedural success | At 12 months after the baseline imaging procedure
  This is the cumulative variable comprising outcomes of each procedure. Ability to complete the imaging procedures without imaging device or procedure related complication.
Change of complexity of coronary artery disease from baseline to follow-up as assessed by SYNTAX score I | At baseline and 12 months after the baseline imaging procedure
  Calculated with the version 2.11 of the SYNTAX Score I calculator at: hospital, at 12 months. The variable will be adjusted for CCTA and QCA due to technical limitations. CT SYNTAX score I will be calculated within recommendations Papadopoulou SL, et al, 2013 (JACC Cardiovasc Imaging. 2013 Mar;6(3):413-5. doi: 10.1016/j.jcmg.2012.09.013; http://www.syntaxscore.com/calculator/syntaxscore/frameset.htm; https://syntaxscore2020.com/).
Change of complexity of coronary artery disease from baseline to follow-up as assessed by SYNTAX score II | At baseline and 12 months after the baseline imaging procedure
  Calculated with the version 2.11 of the SYNTAX Score II calculator at: hospital, at 12 months. The variable will be adjusted for CCTA and QCA due to technical limitations. CT SYNTAX score II will be calculated within recommendations Papadopoulou SL, et al, 2013 (JACC Cardiovasc Imaging. 2013 Mar;6(3):413-5. doi: 10.1016/j.jcmg.2012.09.013; http://www.syntaxscore.com/calculator/syntaxscore/framesetss2.htm; https://syntaxscore2020.com/).
Change of fractional flow reserve (FFR) from baseline to follow-up that are related to the progress of atherosclerosis | At baseline and 12 months after the baseline imaging procedure
  FFR less than 0.75-0.80 considered as hemodynamically significant and estimated for all the lesions. The variable will be adjusted for CCTA and QCA due to technical limitations. FFR will be compared with other variables (QFR of Medis Suite QFR, FFR-CT) including anatomical and functional imaging such as CCTA/ MSCT, CMR, SPECT, OCT, IVUS, VH-IVUS to evaluate any correlations.
Number of participants with contrast-induced nephropathy (CIN) | At baseline and 12 months after the baseline imaging procedure
  This is the cumulative variable comprising outcomes of each procedure. Mehran's criteria for CIN diagnosis (validated at 48-72 hours after exposure of each imaging procedure) as well as CIN risk score will be assessed.
Number of participants with radiocontrast-induced thyroid dysfunction | At baseline and 12 months after the baseline imaging procedure
  The serum thyroid-stimulating hormone (TSH) will be examined as the initial test for screening. In case of the clinical manifestation of the thyroid dysfunction, the concentrations of the serum TSH, thyroid peroxidase (TPO) antibody titers, free thyroxine (T4) and free triiodothyronine (T3) will be assessed.
Safety of QCA and CCTA as assessed by the calculation of effective radiation dose | At 12 months after the baseline imaging procedure
  The cumulative effective radiation dose (mSv), signal, noise, contrast (mean signal-signal in left ventricular myocardium), signal-to-noise ratio (SNR) and contrast-to-noise (CNR) ratio will be compared.
Change of complexity of coronary artery disease from baseline to follow-up as assessed by Leaman Coronary Score | At baseline and 12 months after the baseline imaging procedure
  Calculated within the recommendations of Leaman DM, et al, 1981 (Circulation 63, No. 2, 1981) at: hospital, at 12 months. The variable will be adjusted for CCTA and QCA due to technical limitations. CT-Leaman score will be calculated within the recommendations of Mushtaq S, et al, 2015 (Circ Cardiovasc Imaging. 2015 Feb;8(2):e002332. doi: 10.1161/CIRCIMAGING.114.002332).
Number of participants with encephalopathy | At 12 months after the baseline imaging procedure
  The clinical manifestation (medical history, mental status testing with the mini-mental state examination (MMSE) and mini-cog, a physical and neurological exam) of degenerative and/ or paroxysmal encephalopathy will be evaluated with multi-slice computed tomography (MSCT)-screening of the cerebrovascular disease and Alzheimer's disease in association with markers of Herpes Simplex Virus Type 1 (HSV-1) and fungi.
Number of chest pain patients with non-obstructive coronary artery disease | At 12 months after the baseline imaging procedure
  Patients with the negative acute markers of the myocardial damage (myoglobin, troponin I, CK, CK-MB, NT-proBNP) and without hemodynamically significant (<50% stenosis) coronary atherosclerosis verified by CCTA.
Number of chest pain patients without coronary artery disease | At 12 months after the baseline imaging procedure
  Patients with the negative acute markers of the myocardial damage (myoglobin, troponin I, CK, CK-MB, NT-proBNP) and without coronary atherosclerosis verified by CCTA.
Change of global longitudinal strain | At baseline and 12 months after the baseline imaging procedure
  Global longitudinal strain (GLS) will be assessed by the TTE (transthoracic echocardiogram) and then compared with the data from CMR, CCTA/ MSCT and SPECT. The findings will be examined with the validated software of Medis Suite Ultrasound/ AMID (https://medisimaging.com/ultrasound; http://www.amid.net/). The data of CMR including time signal intensity (TSI), delayed signal intensity (DSI), T1, T2 analysis will be assessed by the Medis Suite MR and compared with TTE data,
Difference of direct effects between two groups with various imaging strategies on cost-effectiveness calculating cost of imaging testing | At 12 months after the baseline imaging procedure
  Cost of imaging testing in both groups will be calculated and compared in U.S. dollars and then matched with cost of complications due to imaging testing, effects of radiation, effects of contrast material, other complications of noninvasive and invasive imaging, psychological effects of the imaging test. The difference between groups will be assessed.
Difference of indirect effects between two groups with various imaging strategies on cost-effectiveness calculating cost of the treatment | At 12 months after the baseline imaging procedure
  Cost of the treatment in both groups will be calculated and compared in U.S. dollars and then matched with cost of complications of treatment, cost of health outcome, medical pathway, and health outcome depending on a medical decision based on the image test result, psychological effects of the test result. The difference between groups will be assessed.
Change of wall shear stress | At baseline and 12 months after the baseline imaging procedure
  The wall shear stress (WSS) will be assessed using the imaging data of CCTA and QCA in both groups in dynamics from baseline to 12-month follow-up. The data of WSS will be compared with other anatomical and functional imaging modalities as well as clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kharlamov, M.D., FESC, FACC, FEACVI, Study Chair — De Haar Research Task Force, Amsterdam-Rotterdam, The Netherlands; Alexey Sozykin, M.D., D.Sc., Study Director — Central Clinical Hospital of the Russian Academy of Sciences
Locations (4):
- De Haar Research Foundation, Tallinn, Estonia
- De Haar Research Task Force, Amsterdam, North Holland, Netherlands
- Russia (2):
  - Center of Endosurgery and Lithotripsy, Moscow, Russia, Moscow
  - Central Clinical Hospital of the Russian Academy of Sciences, Moscow

IPD SHARING:
Plan to Share IPD: Undecided
The specific design of the study makes it infeasible to share the required information with the other researchers. Notwithstanding in case of the scientific inquiries regarding meta-analysis the situation might be considered.

REFERENCES:
- See also: Center of Endosurgery and Lithotripsy, Moscow, Russia — https://www.celt.ru/depart/cardio/
- See also: De Haar Research Task Force/ DHRF (aka De Haar Research Foundation) — https://www.dhrfpro.com/
- See also: Central Clinical Hospital of the Russian Academy of Sciences/ CCH RAS — https://www.ckbran.ru/en/
- See also: Medis Medical Imaging Systems B.V. — https://medisimaging.com/
- See also: Pie Medical Imaging B.V. — https://www.piemedicalimaging.com/
- See also: ElucidVivo Research Edition — https://elucidvivo.com/